CLINICAL TRIAL: NCT02051283
Title: Value of Pretreatment MRI Determined Parameters for Predicting Outcome After Radio-frequency Ablation of Hepatocellular Carcinoma
Brief Title: Pretreatment MRI Predicting Outcome After Radio-frequency Ablation of HCC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: Sbis
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; RFA; MRI
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with HCC eligible for RFA: patients with HCC eligible for RFA
  Interventions: Other: RFA

INTERVENTIONS:
Other: RFA — RFA

SUMMARY:
HCC is classified as keratin (K) 19 positive or K19 negative. K19 is a biliary/hepatic progenitor cell (HPC) marker only expressed in a subset of HCC with poor prognosis and high risk of early recurrence after treatment; particularly in radio-frequency ablation (RFA). These patients consequently show worse survival compared to patients with K19 negative HCC.

A recent publication has shown the value of pretreatment biopsy with K19 staining and suggests that the role of routine biopsies in potentially curable HCC should be reconsidered.

However, currently, pretreatment biopsies are rarely performed in the diagnosis of HCC due to the excellent performance of magnetic resonance imaging (MRI) in detection, diagnosis and staging of cirrhotic livers.

Previous publications have indicated imaging patterns that may be associated with worse prognostic tumoral parameters.

If MRI determined imaging parameters could indeed provide a surrogate marker for presence of K19 and/or microvascular invasion as potential important prognostic factors in RFA of HCC, these imaging parameters may thus hold prognostic information towards RFA treatment and possibly predict treatment outcome. .

The purpose of the retrospective study is thus to evaluate MRI determined imaging parameters at pretreatment MRI for their predictive value towards outcome (disease free survival) of radio-frequency ablation for hepatocellular carcinoma.

If successful, pretreatment MRI parameters may be used for selecting patient with high risk of unfavorable outcome after RFA and select the patients for more aggressive treatment such as surgical resection or upfront transplantation.

DETAILED DESCRIPTION:
Recent pathological, immunohistochemical and molecular profiling have progressively revealed the complex classification of primary liver cancers and have resulted in a subclassification roughly separating mucinous cholangiocarcinomas from mixed tumors from "pure" hepatocellular carcinoma (HCC).

In addition, HCC is classified as keratin (K) 19 positive or K19 negative. K19 is a biliary/hepatic progenitor cell (HPC) marker only expressed in a subset of HCC with poor prognosis and high risk of early recurrence after treatment; particularly in radio-frequency ablation (RFA). These patients consequently show worse survival compared to patients with K19 negative HCC.

A recent publication has shown the value of pretreatment biopsy with K19 staining and suggests that the role of routine biopsies in potentially curable HCC should be reconsidered.

However, currently, pretreatment biopsies are rarely performed in the diagnosis of HCC due to the excellent performance of magnetic resonance imaging (MRI) in detection, diagnosis and staging of cirrhotic livers. This progression of MRI is based on technical refining of three-phase contrast-enhanced imaging, development of the cellular marker sequence diffusion-weighted MRI (DWI) and hepatospecific biliary contrast-agents. While pretreatment biopsies would have incremental value in treatment planning, its routine application in daily clinical practice is faced with multiple problems. First, K19 evaluation at histopathology can - in most cases - only reliably be performed on whole resection specimens and is more difficult on biopsies. Second, routine biopsies would lead to a dramatic increase in workload for radiologists and pathologists influencing daily practice and organization. Also, lesions are not always readily detectable at ultrasound and possibly not eligible for percutaneous biopsy requiring laparoscopy guided biopsy under anesthesia. Third, the risk of tract seeding remains controversial but has not been completely excluded.

Previous publications have indicated imaging patterns that may be associated with worse prognostic tumoral parameters. The corona sign seen at CT during arterial portography and hepatic arteriography (invasive imaging only performed in Japan) is associated with the presence of microvascular invasion. However, this sign has not yet been described at MRI. Also MRI derived parameters may predict the presence of HCC expressing progenitor cell markers, including K19. If MRI determined imaging parameters could indeed provide a surrogate marker for presence of K19 and/or microvascular invasion as potential important prognostic factors in RFA of HCC, these imaging parameters may thus hold prognostic information towards RFA treatment and possibly predict treatment outcome. The hypothesis is that lesions showing features correlating to K19 positivity such as persistent (rim) enhancement and rim like intensity at DWI may correlate to worse prognosis than HCC that don't express these imaging features.

If confirmed, MRI may be the first line modality adapting the patients management; either by selecting patients who actually would benefit from biopsy or identifying patients in who more invasive treatment is necessary (for instance: surgical resection instead of RFA in child A patients; ablation with wider margins in patients not eligible for surgery).

However, before performing a prospective or interventional study, experience needs to be gained with the various possible imaging patterns, aiming to find significant correlations between imaging parameters and adverse prognosis.

The purpose of the retrospective study is thus to evaluate MRI determined imaging parameters at pretreatment MRI for their predictive value towards outcome (disease free survival) of radio-frequency ablation for hepatocellular carcinoma.

If successful, pretreatment MRI parameters may be used for selecting patient with high risk of unfavorable outcome after RFA and select the patients for more aggressive treatment such as surgical resection or upfront transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Documented and diagnosed liver confined hepatocellular carcinoma by existing imaging criteria according to currently accepted international guidelines (< 4cm).
* Treatment radio-frequency ablation - (percutaneous, laparascopy, laparatomy)
* Availability of pretreatment MRI with three phase contrast enhanced images and diffusion-weighted sequence prior to treatment.
* Follow-up of at least 2 years.

Exclusion Criteria:

* Non availability of pathologic confirmation or biopsy during radio-frequency ablation.
* Post-treatment follow-up < 2 years.
* Treatment other than RFA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Documented and diagnosed liver confined hepatocellular carcinoma by existing imaging criteria according to currently accepted international guidelines (< 4cm).
  * Treatment radio-frequency ablation - (percutaneous, laparascopy, laparatomy)
  * Availability of pretreatment MRI with three phase contrast enhanced images and diffusion-weighted sequence prior to treatment.
  * Follow-up of at least 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Predictive value of MRI determined contrast-enhanced and diffusion-weighted sequence pattern towards outcome (tumour recurrence < 1 year versus > 1 year) | 2 years
  Predictive value of MRI determined contrast-enhanced and diffusion-weighted sequence pattern towards outcome (tumour recurrence < 1 year versus > 1 year)

SECONDARY OUTCOMES:
Correlation of predictive MRI parameters with histology obtained from biopsy during radio-frequency ablation (tumor grade, microvascular invasion, Keratin 19 status) | 2 years
  Correlation of predictive MRI parameters with histology obtained from biopsy during radio-frequency ablation (tumor grade, microvascular invasion, Keratin 19 status)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals UZ Leuven, Gasthuisberg, Leuven, Vlaams-Brabant, Belgium